CLINICAL TRIAL: NCT03851003
Title: The Influence of Endometrial Suturing During Cesarean Section on the Risk to Develop Uterine Scar Defect: A Randomized Control Study
Brief Title: The Influence of Endometrial Suturing on the Risk of Uterine Scar Defect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5822-18-SMC
Record Dates: First submitted 2019-02-12; First posted 2019-02-22 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Cesarean Wound Disruption
Keywords: cesarean section; niche; uterine scar defect
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Uterine incision repair will include or exclude suturing of the endometrium
Who Masked: Participant
Masking Description: Women will not know which arm they were allocated to
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometrial suturing (Experimental): Uterine incision repair including suturing of the endometrium
  Interventions: Procedure: Endometrial suturing; Device: Vaginal ultrasonography; Other: Questionnaire
- Non - Endometrial suturing (Experimental): Uterine incision repair without suturing of the endometrium
  Interventions: Procedure: Non- endometrial suturing; Device: Vaginal ultrasonography; Other: Questionnaire

INTERVENTIONS:
Procedure: Endometrial suturing — Suturing will include endometrium during cesarean incision repair
  Arms: Endometrial suturing
Procedure: Non- endometrial suturing — Suturing will not include endometrium during cesarean incision repair
  Arms: Non - Endometrial suturing
Device: Vaginal ultrasonography — All women will be invited six month post operation for vaginal sonographic evaluation of the uterine scar
Other: Questionnaire — All women will be invited six month post operation for filling questionnaire concerning possibility of uterine scar defect ( spotting, pelvic pain, fertility abnormalities )

SUMMARY:
Caesarean section (CS) is the commonest major operation performed on women worldwide with progressively rising incidence. Consequently, long-term adverse sequelae due to uterine scar defect have been increasing. Given the association between uterine scar defect and gynecological symptoms, obstetric complications and potentially with subfertility, it is important to elucidate the etiology in order to develop preventive strategies. Surgical technique of uterine incision closure seems to be the most important determinant of defect formation. The aim of this prospective randomized study is to evaluate specifically the influence of inclusion versus exclusion of the endometrium during suturing the uterine incision on the risk to develop uterine scar defect.

DETAILED DESCRIPTION:
Caesarean section (CS) is the commonest major operation performed on women worldwide with progressively rising incidence. Consequently, long-term adverse sequelae due to uterine scar defect have been increasing. Common gynecological complains include chronic pelvic pain, dyspareunia, dysmenorrhea and postmenstrual spotting and infertility. Obstetric sequelae seem to be increasing such as cesarean scar ectopic pregnancy, placenta previa, and placenta accrete, all associated with major maternal morbidity and even mortality. Given the association between uterine scar defect and gynecological symptoms, obstetric complications and potentially with subfertility, it is important to elucidate the etiology in order to develop preventive strategies. Probable risk factors suggested are single-layer myometrium closure, multiple CSs and uterine retroflexion, however, surgical technique of uterine incision closure seems to be the most important determinant of defect formation. It is proposed that continuous, non-locking absorbable sutures in two layers, without including much of decidua and without undue tight (constricting) pulling of sutures are likely to result in good healing of uterine scar. The aim of this prospective randomized study is to evaluate specifically the influence of inclusion versus exclusion of the endometrium during suturing the uterine incision on the risk to develop uterine scar defect.

Material and Methods Prospective randomized single blinded study conducted in a single tertiary center. All women at term (≥37 weeks of gestation) with singleton pregnancy that are about to go threw cesarean section attending the pre- operative clinics, will be offered to participate in the study. After signing informed consent, women will be block randomized for one of two groups: A- uterine incision repair including suturing of the endometrium, B - uterine incision repair without including the endometrium. All operation will be performed by a single highly skilled obstetrician. All other stages of operations will be similar in both of the groups including: low segment incision, delivery of the fetus and the placenta, uterine revision, intraperitoneal uterine repair, use of stratafix thread in double layer suturing. Operative and post operative data will be collected from the medical files including: operation duration, estimated blood loss, operation complications ( hypotension, bladder gut or vascular perforation ) , post operative complications ( hemorrhage, endometritis, vascular - thromboembolic event, ileus ). All women will be invited to the gynecologic clinics six month post operation for vaginal sonographic evaluation of the uterine scar and for filling questionnaire concerning possibility of uterine scar defect ( spotting, pelvic pain, fertility abnormalities ).

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy (≥37 weeks of gestation)
* Elective CS

Exclusion Criteria:

* Uterine scar
* Thrombophilia
* Dysmorphic uterus
* Connective tissue disorder

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 130 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with uterine scar defect six month post cesarean section | Until six month post cesarean section, and through study completion, an average of 1 year
  Uterine scar defect with residual myometrium thickness of less then 2.5 mm

SECONDARY OUTCOMES:
Spotting | Through study completion, an average of 1 year
  The rate of spotting complains since operation reported by the women
Abdominal pain | Through study completion, an average of 1 year
  The rate of abdominal pain since operation reported by the women and estimated by "The Visual Analogue Scale" (VAS) for the estimation of pain. In this scale, women will be asked to mark the pain that they are experiencing on a 10cm-long horizontal line labeled "no pain" on the far left and "worst pain ever" on the far right. Pain intensity is determined by the length of the line as measured from the left-hand side to the point marked. The following cut points on the pain VAS will be use: no pain (0-0.4 cm), mild pain (0.5-4.4 cm), moderate pain (4.5-7.4 cm), and severe pain (7.5-10 cm).

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Aya Mohr-Sasson, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mathai M, Hofmeyr GJ, Mathai NE. Abdominal surgical incisions for caesarean section. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD004453. doi: 10.1002/14651858.CD004453.pub3. PMID 23728648
- [Result] Wang CB, Chiu WW, Lee CY, Sun YL, Lin YH, Tseng CJ. Cesarean scar defect: correlation between Cesarean section number, defect size, clinical symptoms and uterine position. Ultrasound Obstet Gynecol. 2009 Jul;34(1):85-9. doi: 10.1002/uog.6405. PMID 19565535
- [Result] Tulandi T, Cohen A. Emerging Manifestations of Cesarean Scar Defect in Reproductive-aged Women. J Minim Invasive Gynecol. 2016 Sep-Oct;23(6):893-902. doi: 10.1016/j.jmig.2016.06.020. Epub 2016 Jul 5. PMID 27393285
- [Result] van der Voet LF, Bij de Vaate AM, Veersema S, Brolmann HA, Huirne JA. Long-term complications of caesarean section. The niche in the scar: a prospective cohort study on niche prevalence and its relation to abnormal uterine bleeding. BJOG. 2014 Jan;121(2):236-44. doi: 10.1111/1471-0528.12542. PMID 24373597
- [Result] Sholapurkar SL. Etiology of Cesarean Uterine Scar Defect (Niche): Detailed Critical Analysis of Hypotheses and Prevention Strategies and Peritoneal Closure Debate. J Clin Med Res. 2018 Mar;10(3):166-173. doi: 10.14740/jocmr3271w. Epub 2018 Jan 26. PMID 29416572
- [Result] Vervoort AJ, Uittenbogaard LB, Hehenkamp WJ, Brolmann HA, Mol BW, Huirne JA. Why do niches develop in Caesarean uterine scars? Hypotheses on the aetiology of niche development. Hum Reprod. 2015 Dec;30(12):2695-702. doi: 10.1093/humrep/dev240. Epub 2015 Sep 25. PMID 26409016